CLINICAL TRIAL: NCT02671604
Title: Is Rhabdomyolysis an Anesthetic Complication in Patients Undergoing Robot-assisted Radical Prostatectomy?
Brief Title: Rhabdomyolysis and Robot-assisted Radical Prostatectomy
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulsah Karaoren, MD, Umraniye Education and Research Hospital
Other Study IDs: GK9
Record Dates: First submitted 2016-01-21; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Rhabdomyolysis
Keywords: acute renal failure; prostatectomy; minimal invasive surgery
MeSH Terms: conditions — Rhabdomyolysis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
In patients undergoing robot-assisted radical prostatectomy (RARP), pneumoperitoneum, intraoperative fluid restriction and prolonged Trendelenburg position may cause rhabdomyolysis (RM) due to hypoperfusion in gluteal muscles and lower extremities.

In this study, it was aimed to assess effects of BMI, comorbidities, intraoperative positioning, fluid restriction and length of surgery on development of RM in RARP patients during perioperative period.

DETAILED DESCRIPTION:
Fifty-two ASA I-II patients aged 50-80 years, BMI >25 kg/m2 scheduled for an elective RARP were enrolled to the study.

In all patients, pre-anesthetic evaluations including laboratory tests and Charlson Comorbidity Index (CCI) were performed one week before surgery in anesthesia clinic. Comorbid diseases were rated based on CCI. A 4-points scale was used to rate comorbid conditions [1 mild; 4 severe]. Comorbidity grading was performed by adding scores given for each comorbid disease. Based on the grading, patients were stratified into 4 groups as follows: grade 0, 1-2, 3-4 and ≥ 5

In the operation room, intubation was performed after standard anesthesia For surgery, patients were placed in low lithotomy position. All patients were placed on a soft sponge mattress and soft padding gel pads were provided above the shoulders. The patients were placed in a 30-degree STP after achieving pneumoperitoneum at an intra-abdominal pressure level of 15 mmHg. After placing patient to desired position (T0), blood samples were drawn for measurements of ABG, Na, Cl, Ca, K, BUN, Cr, AST, ALT, LDH, cTp-I, CK-MB and CPK.

During the operation, normal saline (1 m/kg/hr) and 6% HES 200/05 (1 ml/kg/hr) infusions were applied. Operation time (OT) and Trendelenburg time (TT) were recorded in all patients.

Blood samples were repeated on the hours 6 (T6), 12 (T12) and 24 (T24) after beginning of surgery. Hydration with 2000 ml crystalloid solution was given until hour 24 after surgery. In all patients, urine output was monitored.

Rhabdomyolysis was defined as postoperative serum CPK level exceeding 5,000 IU/L. It was planned to manage these patients with hypervolemic therapy, correction of acidosis by using IV sodium bicarbonate and stimulation of diuresis by IV furosemide with a goal of maintaining minimal diuresis of 60 ml/hr at pH level of 7.

Postoperative RF was defined as an increase in serum creatinine of 1mg/dl/day (or 90 mmol/l/day) for 2 consecutive days beyond the baseline.

Patients were discharged with control laboratory tests, including the same parameters, on the hour 48 (T48) postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Aged 50-80 years,
* BMI >25 kg/m2
* Patients scheduled for an elective RARP

Exclusion Criteria:

* Patients with ASA III-IV risk status,
* Patients with comorbid diseases that can cause increased muscular activity such as severe dystonia or status asthmaticus,
* Patients with renal or hepatic failure and patients on statin or steroid therapy were excluded.
* Patients converted to laparotomy during surgery.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients scheduled for an elective Robot assisted radical prostatectomy were enrolled to the study.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With serumCreatine Phosphokinase Values greater than 5000IU/L | Change from Baseline Creatine Phosphokinase at 24 hours.
  Rhabdomyolysis was defined as postoperative serum Creatine Phosphokinase level exceeding 5000 IU/L.

SECONDARY OUTCOMES:
number of patients with abnormal laboratory values | on the hours 0 (T9), 6 (T6), 12 (T12) and 24 (T24) after beginning of surgery.
  Laboratory values of serum Na, Cl, Ca, K, BUN, Cr, AST, ALT, LDH, cTp-I, CK-MB

CONTACTS AND LOCATIONS:
Overall Officials: eyup v kucuk, md, Study Director — Umraniye Education and Research Hospital
Locations (1):
- gulsah Karaoren, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim TK, Yoon JR, Lee MH. Rhabdomyolysis after laparoscopic radical nephrectomy -A case report-. Korean J Anesthesiol. 2010 Dec;59 Suppl(Suppl):S41-4. doi: 10.4097/kjae.2010.59.S.S41. Epub 2010 Dec 31. PMID 21286457
- [Result] Vijay MK, Vijay P, Kundu AK. Rhabdomyolysis and myogloginuric acute renal failure in the lithotomy/exaggerated lithotomy position of urogenital surgeries. Urol Ann. 2011 Sep;3(3):147-50. doi: 10.4103/0974-7796.84965. PMID 21976928